CLINICAL TRIAL: NCT02647372
Title: Deep Brain Stimulation for the Treatment of Parkinson's Disease: Comparative Analysis of Clinical Effect of Stimulation of the Globus Pallidus Internus and Subthalamic Nucleus
Brief Title: Deep Brain Stimulation for Parkinson's Disease: the Globus Pallidus Internus Versus Subthalamic Nucleus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Erich Fonoff, MD, PhD, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSL 2012/12
Record Dates: First submitted 2015-11-10; First posted 2016-01-06 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Parkinson Disease
Keywords: parkinson; deep brain stimulation; globus pallidus; subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endocrinological approach (Experimental): Parkinson patient submitted to DBS surgery target to globus pallidus nucleus or the subthalamic nucleus. Those patients will be endocrinological evaluation including metabolic measures, calorimetric parameters.
  Interventions: Procedure: Subthalamic nucleus; Procedure: Globus pallidus
- Neurological approach (Experimental): Parkinson patient submitted to DBS surgery target to globus pallidus nucleus or the subthalamic nucleus. Those patients will be neurological evaluation including UPDRS scale.
  Interventions: Procedure: Subthalamic nucleus; Procedure: Globus pallidus

INTERVENTIONS:
Procedure: Subthalamic nucleus — Surgery will be performed in 15 patients with DBS target to the subthalamic nucleus
Procedure: Globus pallidus — Surgery will be performed in 15 patients with DBS target to the globus pallidus nucleus

SUMMARY:
This study provides an evaluation of 30 patients in 3 years, from the Unified Health System (SUS) irrespective of region of the country, signed with clinical Parkinson's disease in its intermediate stage and that the drug therapy is limited by side effects or beneficial effects provided by prior medication no longer be obtained even at high doses and have therefore the indication for treatment with deep brain stimulation.

DETAILED DESCRIPTION:
The aim of this retrospective study is to compare motor and non-motor (olfactory, pain, cognition and metabolism) symptoms of the effects of deep brain stimulation target to the nucleus globus pallidus versus the subthalamic nucleus in patients with Parkinson´s disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of idiopathic Parkinson's disease according to the international criteria that have not responded adequately to treatment with medication or who have complications related to prolonged use of L-dopa.
* Patients who may be in the anesthetized or local or general anesthesia does not incur higher than expected risk in the general population.
* Patients intellectually able to understand and sign the consent form.
* Patients with hematological, metabolic and normal coagulation.

Exclusion Criteria:

* Age below 18 years
* Impossibility to consent to participate in the study.
* Patients during treatment with anti-coagulants or anti-platelet agents.
* Patients with anatomical abnormalities that preclude access to the implantation of electrodes (eg cranial tumors or intracranial or cysts).
* Patients with uncontrolled infection or other medical conditions pre-existing non-controlled (eg decompensated diabetes, hypertension, heart disease or symptomatic air).
* History of primary or secondary myocardial ischemia, congestive heart failure, cardiac arrhythmia or bundle branch block refractory to treatment.
* Concomitant treatment with other experimental drugs.
* Pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Neurological approach measured by UPDRS scale | through study completion, an average of 2 years
  UPDRS scale before surgery
Neurological approach measured by UPDRS scale | 6 months
  UPDRS scale 6 months after surgery
Neurological approach measured by UPDRS scale | 12 months
  UPDRS scale 12 months after surgery
Neurological approach measured by UPDRS scale | 24 months
  UPDRS scale 24 months after surgery

SECONDARY OUTCOMES:
Endocrinological approach | through study completion, an average of 2 years
  Evaluation of metabolic measures before surgery
Endocrinological approach | 6 months
  Evaluation of metabolic measures 6 months after surgery
Endocrinological approach | 12 months
  Evaluation of metabolic measures 12 months after surgery
Endocrinological approach | 24 months
  Evaluation of metabolic measures 24 months after surgery
Endocrinological approach - BMI | 36 months
  Evaluation of body mass index before surgery
Endocrinological approach - BMI | 6 months
  Evaluation of body mass index 6 months after surgery
Endocrinological approach - BMI | 12 months
  Evaluation of body mass index12 months after surgery
Endocrinological approach - BMI | 24 months
  Evaluation of body mass index 24 months after surgery